CLINICAL TRIAL: NCT01567384
Title: A Phase I Study of OSI-906 in Combination With Pemetrexed in Advanced Solid Tumor Malignancies
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: The sponsor withdrew support for the study before any patients were enrolled.
Sponsor: Emory University (Other)
Collaborators: OSI Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Suresh S. Ramalingam, Principal Investigator, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00047570; WCI1895-10 (Other: Other)
Record Dates: First submitted 2011-12-20; First posted 2012-03-30 (Estimated); Last update posted 2013-11-20 (Estimated); Status verified 2013-11

CONDITIONS: Cancer; Neoplasms; Tumors
Keywords: cancer; neoplasms; tumors
MeSH Terms: conditions — Neoplasms | interventions — 3-(8-amino-1-(2-phenylquinolin-7-yl)imidazo(1,5-a)pyrazin-3-yl)-1-methylcyclobutanol; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Combination therapy with OSI and Pemetrexed (Experimental)
  Interventions: Drug: OSI-906 and Pemetrexed

INTERVENTIONS:
Drug: OSI-906 and Pemetrexed — Pemetrexed will be administered intravenously on day 1 of cycle 1 at a dose of 500 mg/m2 as a 10-minute infusion. Subsequent doses will be defined by tolerability.
  OSI-906 will be administered orally twice daily (12 hours apart) at approximately the same times each day on a continuous schedule, beginning on Day 0 of cycle 1.

SUMMARY:
The purpose of the study is to test the safety of an experimental drug called OSI-906 when combined with pemetrexed at different dose levels and to find out the optimal doses of the two drugs that can be given as a combination. Pemetrexed has been widely used for treatment of certain solid organ tumors and is effective and approved for use in treatment of lung cancer and mesothelioma.

DETAILED DESCRIPTION:
OSI-906 is a new agent that inhibits the insulin-like growth factor receptor pathway. Targeting this pathway appears to be a promising strategy to treat cancer based on laboratory studies. The present study will test if this agent can be administered safely in combination with pemetrexed, a commonly used chemotherapeutic agent.

ELIGIBILITY:
Inclusion Criteria:

* Both men and women of all races and ethnic groups are eligible for this trial.
* Patients must have histologically confirmed malignancy.
* Patient's tumor type must be appropriate for therapy with pemetrexed or have no standard treatment approaches.
* Patients must have discontinued previous chemotherapy and/or radiation at least 3 weeks[six weeks for nitrosoureas, BCNU, or mitomycin C] prior to entry into the study and recovered from any toxic effects of previous treatment. Pallative radiation therapy to sites involving more than 2 weeks prior to enrollment on this study.
* Age greater than 18 years.
* ECOG performance status less than 2 [see Appendix A].
* Patients should be able to take oral medications.
* Patients must have normal organ and marrow function as defined below:
* leukocytes greater than 3,000/mcL
* absolute neutrophil count greater than 1,500/mcL
* platelets greater than 100,000/mcL
* total bilirubin within normal institutional limits AST[SGOT]/ALT[SGPT]less than 2.5 x institutional upper limit of normal
* creatinine within normal institutional limits OR
* creatinine clearance greater than 60 mL/min/1.73 m2 for patients with creatinine levels above institutional normal.
* The effects of OSI-906 on the developing human fetus are unknown. For this reason and because chemotherapeutic agents as well as other therapeutic agents used in this trial are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception [hormonal or barrier method of birth control; abstinence] prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Patients may not be receiving any other investigational agents.
* Patients with untreated, active or symptomatic brain metastases should be excluded from this clinical trial.
* History of allergic reaction to OSI-906 or pemetrexed.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit adherence with study requirements.
* Pregnant women are excluded from this study because OSI-906 and pemetrexed are anti-proliferative agents agent with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with OSI-906, breastfeeding should be discontinued if the mother is treated OSI-906. These potential risks may also apply to other agents used in this study.
* HIV-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with OSI-906. In addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy. Appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated.
* Patients with QTc interval greater than 450 msec at baseline will be excluded due to risk of QTc prolongation with OSI-906.
* Patients taking medications that prolong the QTc interval will be excluded.
* Patients with significant cardiac disease will be excluded.
* Patients with fasting blood glucose greater than 150 mg/dL at baseline will be excluded due to risk of hyperglycemia with OSI-906.
* Use of drugs that have a known risk of causing Torsades de Pointes [TdP] [Torsades List on www.azcert.org/medical-pros/drug-lists/bycategory.cfm, see Appendix D] are prohibited within 14 days prior to randomization.
* Use of the potent CYP1A2 inhibitors ciprofloxacin and fluvoxamine. Other less potent CYP1A2 inhibitors/inducers are not excluded.
* Patients with a history of poorly controlled gastrointestinal disorders that could affect the absorption of study drug (eg, Crohn's disease, ulcerative colitis, etc) should be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-05; Primary Completion 2013-10 (Estimated); Study Completion 2013-10 (Estimated)

PRIMARY OUTCOMES:
Assessment of dose-limiting toxicity | 21 days
  To define the dose of OSI-906 that can be combined with pemetrexed

SECONDARY OUTCOMES:
Progression-free survival | 4-6 months
  Response and progression will be evaluated in this study using the new international criteria proposed by the revised Response Evaluation Criteria in Solid Tumors (RECIST) guideline (version 1.1) [Eur J Ca 45:228-247, 2009]. Changes in the largest diameter (unidimensional measurement) of the tumor lesions and the shortest diameter in the case of malignant lymph nodes are used in the RECIST criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Suresh Ramalingam, MD, Principal Investigator — Emory University
Locations (1):
- Winship Cancer Institute of Emory University, Atlanta, Georgia, United States